CLINICAL TRIAL: NCT01698099
Title: Diagnostic Accuracy of Serum Bilirubin in the Prediction of Perforated Appendicitis
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Sven Mueller, Principal Investigator, University Hospital Tuebingen
Other Study IDs: APP001
Record Dates: First submitted 2012-09-24; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hyperbilirubinemia is reported to be a positive predictor in diagnosing perforated appendicitis. Therefore we analysed the diagnostic accuracy of serum bilirubin in discriminating between perforated and simple/no appendicitis.

Methods:

All consecutive patients undergoing appendectomy for suspected appendicitis from May 2009 to August 2011 were analysed. Primary endpoint was the diagnostic accuracy of serum bilirubin levels to detect perforated appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing appendectomy for suspected appendicitis

Exclusion Criteria:

* preexisting liver disease

Ages: 16 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing appendectomy for suspected appendicitis
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2009-05; Primary Completion 2011-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of serum bilirubin | 24h within initial presentation with clinical symptoms
  assessment of the diagnostic accuracy of hyperbilirubinemia (defined as serum bilirubin above 1.1 md/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Müller, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- Departement of Visceral- and Transplant Surgery, University of Tuebingen, Tübingen, Germany

REFERENCES:
- [Derived] Muller S, Falch C, Axt S, Wilhelm P, Hein D, Konigsrainer A, Kirschniak A. Diagnostic accuracy of hyperbilirubinaemia in anticipating appendicitis and its severity. Emerg Med J. 2015 Sep;32(9):698-702. doi: 10.1136/emermed-2013-203349. Epub 2014 Dec 4. PMID 25476715